CLINICAL TRIAL: NCT03688100
Title: Personalized Treatments for Depressive Symptoms in Patients With Advanced Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Waguih William IsHak, MD, FAPA, Vice Chair, Education and Research in the Department of Psychiatry and Behavioral Neurosciences, Professor Psychiatry & Behavioral Neurosciences, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00054483
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Results first posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-02

CONDITIONS: Depression; Heart Failure
MeSH Terms: conditions — Depression; Heart Failure | interventions — Medication Therapy Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Patients: Medication Management (MEDS) (Active Comparator): The medication management group will meet with the patient in a one 50 minute in person introductory antidepressant medication treatment session to educate the patient about depression and medication options. Patients will get prescribed a standard of care anti-depressant medication by treating physician, followed by 12 weekly follow up telephone visits, then on a monthly basis for 3 months, and then as needed thereafter.
  Interventions: Drug: Medication Management
- Patients: Behavioral Activation Therapy (BA) (Active Comparator): BA is an evidence-based psychotherapy with more than 25 randomized trials showing effectiveness in depression. The therapy group will consist of an introductory in person 50-minute treatment session, followed by 12 weekly telephone 50-minute outpatient treatment sessions, then 3 monthly telephone 50-minute outpatient maintenance sessions. A typical BA session will last 50 minutes and include a review of the previous session and completed daily monitoring record forms, an in-depth discussion of life areas and value, and verbal reinforcement of activity engagement.
  Interventions: Behavioral: Behavioral Activation Therapy
- Caregivers: Medication Management (MEDS) (No Intervention): Caregivers of patients receiving the the above described Medication Management (MEDS) intervention were monitored for caregiver burden at 3, 6, and 12 months.
- Caregivers: Behavioral Activation Psychotherapy (BA) (No Intervention): Caregivers of patients receiving the the above described Behavioral Activation Psychotherapy (BA) intervention were monitored for caregiver burden at 3, 6, and 12 months.

INTERVENTIONS:
Behavioral: Behavioral Activation Therapy — The therapy group will consist of an introductory in person 50-minute treatment session, followed by 12 weekly telephone 50-minute outpatient treatment sessions, then 3 monthly telephone 50-minute outpatient maintenance sessions. A typical BA session will last 50 minutes and include a review of the previous session and completed daily monitoring record forms, an in-depth discussion of life areas and value, and verbal reinforcement of activity engagement.
  Other Names: BA
  Arms: Patients: Behavioral Activation Therapy (BA)
Drug: Medication Management — Collaborative care model will be used. The medication management group will meet with the patient in a one 50 minute in person introductory antidepressant medication treatment session to educate the patient about depression and medication options. Patients will get prescribed a standard of care anti-depressant medication by treating physician, followed by 12 weekly follow up telephone visits, then on a monthly basis for 3 months, and then as needed thereafter.
  Other Names: MEDS
  Arms: Patients: Medication Management (MEDS)

SUMMARY:
We are doing this study to help patients, caregivers, and providers make decisions about how best to manage depressive symptoms in advanced heart failure. There are two evidence-based treatment approaches to treating depression in patients with advanced heart failure, behavioral action psychotherapy and treatment with anti-depressant medications. In this study we want to compare the effectiveness of these two treatment options to learn which treatment works better.

DETAILED DESCRIPTION:
Aim 1: To compare the effectiveness of BA vs. MEDS, for depressed AHF patients. Hypothesis 1: Compared to depressed AHF patients who receive MEDS, patients receiving BA will have significantly greater improvements in the primary outcome of depressive symptom severity as measured with the PHQ-9 at 6-month follow-up. Significantly greater improvements will also be detected in the secondary outcomes of general physical and mental HRQoL (SF-12v2), heart failure-specific HRQoL (KCCQ), and caregiver burden (CBQ-HF) at 3, 6, and 12 months.

Aim 2: To compare the impact of BA vs. MEDS on disadvantageous outcomes of Morbidity (as evidenced by ED visits, hospital readmissions, total days in the hospital), and Mortality among depressed AHF patients.

Hypothesis 2: Compared to depressed AHF patients who receive MEDS, those receiving BA will have significantly less Morbidity (as evidenced by less frequent ED visits, lower readmission rates, fewer total days in the hospital), and reduced Mortality at the data collection points of 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. HF New York Heart Association classes: II-IV.
2. Life expectancy of more than 6 months.
3. PHQ-9 score ≥10.
4. Diagnosis of Major Depressive Disorder, Persistent Depressive Disorder (Dysthymia), and Depressive Disorder Unspecified, as confirmed by the MINI 7.02.

Exclusion Criteria:

1. Imminent danger to self or others.
2. Cognitive impairments with a MOCA score of < 23.
3. Bipolar, Psychotic, and Substance-induced Disorders.
4. Patients in active treatment of depression who are already on antidepressants, psychotherapy, or both.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2022-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Waguih W IsHak, MD, FAPA, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] IsHak WW, Hamilton MA, Korouri S, Diniz MA, Mirocha J, Hedrick R, Chernoff R, Black JT, Aronow H, Vanle B, Dang J, Edwards G, Darwish T, Messineo G, Collier S, Pasini M, Tessema KK, Harold JG, Ong MK, Spiegel B, Wells K, Danovitch I. Comparative Effectiveness of Psychotherapy vs Antidepressants for Depression in Heart Failure: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jan 2;7(1):e2352094. doi: 10.1001/jamanetworkopen.2023.52094. PMID 38231511
- [Derived] IsHak WW, Korouri S, Darwish T, Vanle B, Dang J, Edwards G, Black JT, Aronow H, Kimchi A, Spiegel B, Hedrick R, Chernoff R, Diniz MA, Mirocha J, Manoukian V, Harold J, Ong MK, Wells K, Hamilton M, Danovitch I. Personalized treatments for depressive symptoms in patients with advanced heart failure: A pragmatic randomized controlled trial. PLoS One. 2021 Jan 7;16(1):e0244453. doi: 10.1371/journal.pone.0244453. eCollection 2021. PMID 33412562

RESULTS

PARTICIPANT FLOW:
Groups:
- Caregivers: Medication Management (MEDS): Caregivers in the medication management group do not participate in the medication management intervention. Rather, the medication management intervention is delivered to patients and the effect of this intervention is on patient's caregivers' burden is measured by the Caregiver Burden Questionnaire.
- Caregivers: Behavioral Activation Psychotherapy (BA): Caregivers in the behavioral activation group do not participate in the behavioral activation intervention. Rather, the behavioral activation intervention is delivered to patients and the effect of this intervention on patient's caregivers' burden is measured by the Caregiver Burden Questionnaire.
Period: Overall Study
Arm/Group | Patients: Medication Management (MEDS) | Patients: Behavioral Activation Therapy (BA) | Caregivers: Medication Management (MEDS) | Caregivers: Behavioral Activation Psychotherapy (BA)
Started | 208 | 208 | 35 | 43
Completed | 132 | 150 | 20 | 25
Not Completed | 76 | 58 | 15 | 18
Not completed — Lost to Follow-up | 21 | 15 | 15 | 18
Not completed — Withdrawal by Subject | 19 | 16 | 0 | 0
Not completed — Death | 36 | 27 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Overall baseline participants include patient participants in each arm, and caregiver participants.
Groups:
- Caregivers: Behavioral Activation Therapy (BA): Caregivers of patients receiving the the above described Behavioral Activation Psychotherapy (BA) intervention were monitored for caregiver burden at 3, 6, and 12 months.
- Total: Total of all reporting groups
Arm/Group | Patients: Medication Management (MEDS) | Patients: Behavioral Activation Therapy (BA) | Caregivers: Medication Management (MEDS) | Caregivers: Behavioral Activation Therapy (BA) | Total
Number analyzed (Participants) | 208 | 208 | 35 | 43 | 494
Age, Continuous [Mean (Standard Deviation); unit: years]
  MEAN AGE | 61 (16) | 61 (16) | 55 (16) | 55 (13) | 61 (16)
Age, Continuous [Median (Inter-Quartile Range); unit: years]
  MEDIAN AGE (IQR) | 61 [51 to 72] | 64 [52 to 71] | 57 [45 to 64] | 59 [45 to 64] | 62 [51 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 88 | 27 | 30 | 230
  Male | 123 | 120 | 8 | 13 | 264
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian/White | 112 | 121 | 19 | 28 | 280
  Race: Black/African-American | 60 | 62 | 6 | 8 | 136
  Race: Asian | 14 | 7 | 2 | 2 | 25
  Race: Other | 22 | 18 | 8 | 5 | 53
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Not Hispanic or Latino | 171 | 173 | 24 | 33 | 401
  Ethnicity: Hispanic or Latino | 32 | 28 | 7 | 9 | 76
  Ethnicity: Missing | 5 | 7 | 4 | 1 | 17
Medications [Number; unit: Number of patients taking the medication]
  Angiotensin Receptor Blocker | 66 | 69 | 0 | 0 | 135
  Loop Diuretic | 142 | 137 | 0 | 0 | 279
  Opiate | 65 | 51 | 0 | 0 | 116
  Angiotensin-Converting Enzyme Inhibitor | 33 | 33 | 0 | 0 | 66
  Beta Blocker | 135 | 133 | 0 | 0 | 268
  Aldosterone Antagonist | 50 | 50 | 0 | 0 | 100
  Calcium Channel Blocker | 48 | 49 | 0 | 0 | 97
  Digoxin | 13 | 25 | 0 | 0 | 38
  Steroid | 39 | 31 | 0 | 0 | 70
  Cannabinoid | 7 | 5 | 0 | 0 | 12
  History of Antidepressant | 60 | 26 | 0 | 0 | 86
  Anticoagulant | 61 | 89 | 0 | 0 | 150
  Ivabradine | 2 | 1 | 0 | 0 | 3
  Non-Loop Diuretic | 3 | 2 | 0 | 0 | 5
  Statin | 110 | 105 | 0 | 0 | 215
  Antiaggregant | 31 | 40 | 0 | 0 | 71
  Antiarrhythmic | 27 | 34 | 0 | 0 | 61
  Angiotensin Receptor Neprilysin Inhibitor | 38 | 38 | 0 | 0 | 76
  Hydralazine and Nitrate | 65 | 58 | 0 | 0 | 123
  Sodium-Glucose-Co-Transporter-2 Inhibitor | 4 | 8 | 0 | 0 | 12
  ACE + ARB + Entresto | 105 | 107 | 0 | 0 | 212
Location of Recruitment [Count of Participants; unit: Participants]
  Inpatient | 107 | 99 | 17 | 22 | 245
  Outpatient | 101 | 109 | 18 | 21 | 249

OUTCOME MEASURES:

1. Primary Outcome: Depressive Symptom Severity as Measured by the Patient Health Questionnaire (PHQ-9) Depression Scale Results at 6 Months Follow up
Description: PHQ-9 is used to measure depressive symptoms severity. The PHQ-9 is a self-report instrument that corresponds with the validated Primary Care Evaluation of Mental Disorders PRIME-MD clinician-administered instrument. The PHQ-9 measures all nine dimensions of depression assessed in the DSM criteria for MDD on a 0-3 scale. Minimum score = 0 (no depression). Maximum scores = 21 (worst depression)
Time Frame: 6 months from baseline enrollment.
Population: Intention-to-treat: We analyzed all participants in both arms who were randomized to their respective intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Medication Management Group: The medication management group will meet with the patient in a one 50 minute in person introductory antidepressant medication treatment session to educate the patient about depression and medication options. Patients will get prescribed a standard of care anti-depressant medication by treating physician, followed by 12 weekly follow up telephone visits, then on a monthly basis for 3 months, and then as needed thereafter.
  Medication Management: Collaborative care model will be used. The medication management group will meet with the patient in a one 50 minute in person introductory antidepressant medication treatment session to educate the patient about depression and medication options. Patients will get prescribed a standard of care anti-depressant medication by treating physician, followed by 12 weekly follow up telephone visits, then on a monthly basis for 3 months, and then as needed thereafter.
- Behavioral Activation Therapy: BA is an evidence-based psychotherapy with more than 25 randomized trials showing effectiveness in depression. The therapy group will consist of an introductory in person 50-minute treatment session, followed by 12 weekly telephone 50-minute outpatient treatment sessions, then 3 monthly telephone 50-minute outpatient maintenance sessions. A typical BA session will last 50 minutes and include a review of the previous session and completed daily monitoring record forms, an in-depth discussion of life areas and value, and verbal reinforcement of activity engagement.
  Behavioral Activation Therapy: The therapy group will consist of an introductory in person 50-minute treatment session, followed by 12 weekly telephone 50-minute outpatient treatment sessions, then 3 monthly telephone 50-minute outpatient maintenance sessions. A typical BA session will last 50 minutes and include a review of the previous session and completed daily monitoring record forms, an in-depth discussion of life areas and value, and verbal reinforcement of activity engagement.
Arm/Group | Medication Management Group | Behavioral Activation Therapy
Number analyzed (Participants) | 208 | 208
score on a scale
  PHQ-9 at Baseline | 14.31 (3.60) | 14.54 (3.45)
  PHQ-9 at 6 months | 8.09 (6.06) | 7.53 (5.74)

2. Secondary Outcome: Change From Baseline in the 12-item Questionnaire Used to Assess Health-related Quality of Life (SF-12v2) Scale Results
Description: The SF-12v2 is a 12-item questionnaire used to assess Health-related Quality of Life (HRQoL) from the patient's perspective. The SF-12v2 consists of 12 questions from the SF-36 that evaluate the same eight health domains: physical function, the role-physical, bodily pain, general health, vitality, social function, the role-emotional, and mental health. The Physical Component Summary (PCS) and Mental Component Summary (MCS) scores are norm-based scores ranging from 0 to 100 calculated from the responses to the 12 questions using scoring software from QualityMetric.com. In the general US population, the mean normal score is 50, with a standard deviation (SD) of 10. Higher scores indicate better outcomes with better HRQoL. Health-related Quality of Life - Physical Health as measured by SF-12 physical component and Health
Time Frame: 3 month, 6 month, and 12 months from baseline enrollment
Population: Intention to treat: We analyzed all participants in both arms who were randomized to their respective intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients: Medication Management (MEDS) | Patients: Behavioral Activation Therapy (BA)
Number analyzed (Participants) | 208 | 208
score on a scale
  SF-12v2 Physical Component Score at Baseline | 35.56 (7.74) | 35.89 (9.26)
  SF-12v2 Physical Component Score at 3-months | 37.46 (10.17) | 37.69 (10.60)
  SF-12v2 Physical Component Score at 6-months | 37.12 (10.99) | 38.82 (11.09)
  SF-12v2 Physical Component Score at 12-months | 37.72 (10.81) | 37.89 (11.74)
  SF-12v2 MentalComponent Score at Baseline | 37.22 (9.23) | 36.87 (9.16)
  SF-12v2 Mental Component Score at 3-months | 47.63 (10.77) | 48.25 (11.08)
  SF-12v2 Mental Component Score at 6-months | 46.85 (12.55) | 47.33 (10.97)
  SF-12v2 Mental Component Score at 12-months | 47.41 (12.07) | 47.04 (9.91)

3. Secondary Outcome: Change From Baseline on the Kansas City Cardiomyopathy Questionnaire (KCCQ ) Scale Results.
Description: The KCCQ is a 23-item, self-administered instrument that quantifies 6 domains and yields 2 summary scores. The 6 domains are physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. The 2 summary scores are the Clinical Summary Score and the Overall Summary Score. The Clinical Summary score includes total symptom and physical function scores to correspond with NYHA Classification. The Overall Summary Score includes the total symptom, physical function, social limitations and quality of life scores. Domain scores and summary scores are scaled from the raw item scores using a software available from the authors (SPERTUSJ@UMKC.EDU) to a range from 0 (worst) to 100 (best), in which higher scores reflect better heart-failure-specific quality of life and health status. Heart failure-specific quality of life are measured by the KCCQ Overall Summary Score and the Clinical Summary Score .
Time Frame: 3 month, 6 month, and 12 months from baseline enrollment
Population: Intention to treat: We analyzed all participants in both arms who were randomized to their respective intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients: Medication Management (MEDS) | Patients: Behavioral Activation Therapy (BA)
Number analyzed (Participants) | 208 | 208
score on a scale
  KCCQ Overall Summary Score at 3-months | 60.57 (23.03) | 62.03 (25.69)
  KCCQ Overall Summary Score at 6-months | 61.43 (24.48) | 64.35 (26.89)
  KCCQ Overall Summary Score at 12-months | 65.48 (24.83) | 63.24 (25.88)
  KCCQ Clinical Summary Score at 3-months | 64.16 (24.88) | 64.01 (26.76)
  KCCQ Clinical Summary Score at 6-months | 63.39 (25.92) | 66.15 (27.17)
  KCCQ Clinical Summary Score at 12-months | 67.02 (24.43) | 64.00 (27.19)

4. Secondary Outcome: Change From Baseline on the Caregiver Burden Questionnaire-Heart Failure (CBQ-HF) Scale Results.
Description: The Caregiver Burden Questionnaire - Heart Failure Version 3.0 (CBQ-HF) is a quantitative survey of 26 questions covering the past four weeks of the caregiver's experience is evaluated as caregiver burden. The scale uses a 5-point Likert severity scale (Not at all=0, A little=1, Somewhat=2, Quite a lot=3, A lot=4) assessing 4 domains of physical, emotional/psychological, social and lifestyle burdens. The score is summed from all the questions for each domain, and then summed to a total score that ranges from 0 (no burden) to 104 (worst burden), in which higher scores reflect worse outcomes of higher burden on the caregiver. We will measure the caregiver burden measured by the CBQ-HF.
Time Frame: 3 month, 6 month, and 12 months from baseline enrollment
Population: The number analyzed in each row differs from the overall number analyzed because of missing caregiver questionnaire data at each timepoint of 3-months, 6-months, and 12-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregivers: Medication Management (MEDS) | Caregivers: Behavioral Activation Psychotherapy (BA)
Number analyzed (Participants) | 35 | 43
score on a scale
  CBQ-HF Overall Score at Baseline | 68.06 (20.04) | 65.14 (20.96)
  CBQ-HF Overall Score at 3-months: number analyzed (Participants) | 25 | 24
  CBQ-HF Overall Score at 3-months | 61.52 (19.72) | 57.70 (21.62)
  CBQ-HF Overall Score at 6-months: number analyzed (Participants) | 19 | 25
  CBQ-HF Overall Score at 6-months | 57.38 (17.96) | 55.27 (18.13)
  CBQ-HF Overall Score at 12-months: number analyzed (Participants) | 19 | 23
  CBQ-HF Overall Score at 12-months | 63.19 (23.63) | 60.39 (24.98)

5. Secondary Outcome: Mean Number of Emergency Department Visits
Description: We recorded the number of emergency department visits.
Time Frame: 3 month, 6 month, and 12 months from baseline enrollment
Population: Using a Zero Inflated Poisson (ZIP) Model, at 3, 6, and 12 months, the mean ratios of ED visits were compared for patients with heart failure who received BA to those who received MEDS.
Measure: Mean (Full Range); unit: Mean ED visits
Arm/Group | Patients: Medication Management (MEDS) | Patients: Behavioral Activation Therapy (BA)
Number analyzed (Participants) | 208 | 208
Mean ED visits
  Mean ED visits at 3-months | 0.90 [0 to 1] | 0.55 [0 to 1]
  Mean ED visits at 6-months | 1.51 [0 to 2] | 1.31 [0 to 2]
  Means ED visits at 12-months | 2.43 [0 to 3] | 1.87 [0 to 3]
Statistical Analysis 1: Comparison: Patients: Medication Management (MEDS) vs Patients: Behavioral Activation Therapy (BA); Emergency Department visits AT 3 MONTHS; Test type: Superiority; p = 0.005, Zero Inflated Poisson (ZIP) Model — The a priori threshold for statistical significance is p<0.05; ratio of means = 0.62, 95% CI 2-sided [0.45 to 0.86] — For the ratio of means, BA is the numerator and MEDS is the denominator
Statistical Analysis 2: Comparison: Patients: Medication Management (MEDS) vs Patients: Behavioral Activation Therapy (BA); Emergency Department visits AT 6 MONTHS; Test type: Superiority; p = 0.008, Zero Inflated Poisson (ZIP) Model — The a priori threshold for statistical significance is p<0.05; ratio of means = 0.70, 95% CI 2-sided [0.60 to 0.86] — For the ratio of means for ED visits, BA is the numerator and MEDS is the denominator
Statistical Analysis 3: Comparison: Patients: Medication Management (MEDS) vs Patients: Behavioral Activation Therapy (BA); Emergency Department visits AT 12 MONTHS; Test type: Superiority; p = 0.0001, Zero Inflated Poisson (ZIP) Model — The a priori threshold for statistical significance is p<0.05; ratio of means = 0.73, 95% CI 2-sided [0.62 to 0.85] — For the ratio of means for ED visits , BA is numerator and MEDS is the denominator

6. Secondary Outcome: Mean Number of Readmissions (Hospitalization)
Description: We recorded the number of readmissions to the hospital.
Time Frame: 3 month, 6 month, and 12 months from baseline enrollment
Population: Using a Zero Inflated Poisson (ZIP) Model, at 3, 6, and 12 months, the mean ratios of Hospital Admissions were compared for patients with heart failure who received BA to those who received MEDS.
Measure: Mean (Full Range); unit: Mean Hospital Readmissions
Arm/Group | Patients: Medication Management (MEDS) | Patients: Behavioral Activation Therapy (BA)
Number analyzed (Participants) | 208 | 208
Mean Hospital Readmissions
  Mean Hospital Readmissions at 3-months | 0.86 [0 to 1] | 0.67 [0 to 1]
  Mean Hospital Readmissions at 6-months | 1.48 [0 to 2] | 1.30 [0 to 2]
  Mean Hospital Readmissions at 12-months | 2.20 [0 to 3] | 2.00 [0 to 3]
Statistical Analysis 1: Comparison: Patients: Medication Management (MEDS) vs Patients: Behavioral Activation Therapy (BA); Differences in the number of hospital readmissions between BA and MEDS at 3, 6, and 12 months; Test type: Superiority; p > 0.05, Zero Inflated Poisson (ZIP) Model — The a priori threshold for statistical significance is p<0.05

7. Secondary Outcome: If Hospitalized, Mean Number of Total Days in the Hospital
Description: We recorded the number of total days in the hospital if they were hospitalized.
Time Frame: 3 month, 6 month, and 12 months from baseline enrollment
Population: Using a Zero Inflated Poisson (ZIP) Model, the ratio of means were compared for total days in the hospital for BA vs. MEDS, at 3, 6, and 12 months respectively.
Measure: Mean (Full Range); unit: Mean Number ofTotal Days in the Hospital
Arm/Group | Patients: Medication Management (MEDS) | Patients: Behavioral Activation Therapy (BA)
Number analyzed (Participants) | 208 | 208
Mean Number ofTotal Days in the Hospital
  Mean Number of Total Days in the Hospital at 3-months | 5.50 [0 to 6] | 3.84 [0 to 6]
  Mean Number of Total Days in the Hospital at 6-months | 8.79 [0 to 9] | 7.18 [0 to 9]
  Mean Number of Total Days in the Hospital at 12-months | 15.19 [0 to 16] | 11.11 [0 to 16]
Statistical Analysis 1: Comparison: Patients: Medication Management (MEDS) vs Patients: Behavioral Activation Therapy (BA); Days in the Hospital at 3 months; Test type: Superiority; p = 0.002, Zero Inflated Poisson (ZIP) Model — The a priori threshold for statistical significance is p<0.05; ratio of means = 0.83, 95% CI 2-sided [0.75 to 0.92] — For the ratio of means, BA is the numerator and MEDS is the denominator
Statistical Analysis 2: Comparison: Patients: Medication Management (MEDS) vs Patients: Behavioral Activation Therapy (BA); Days in the Hospital at 6 MONTHS; Test type: Superiority; p = 0.005, Zero Inflated Poisson (ZIP) Model — The a priori threshold for statistical significance is p<0.05; ratio of means = 0.81, 95% CI 2-sided [0.75 to 0.87] — For the ratio of means, BA is numerator and MEDS is the denominator
Statistical Analysis 3: Comparison: Patients: Medication Management (MEDS) vs Patients: Behavioral Activation Therapy (BA); Days in the Hospital AT 12 MONTHS; Test type: Superiority; p < 0.0001, Zero Inflated Poisson (ZIP) Model — The a priori threshold for statistical significance is p<0.05; ratio of means = 0.64, 95% CI 2-sided [0.60 to 0.68] — For the ratio of means, BA is the numerator and MEDS is the denominator

8. Secondary Outcome: Mortality Was Also Measured
Description: We recorded mortality data on the patients.
Time Frame: 3 month, 6 month, and 12 months from baseline enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Patients: Medication Management (MEDS) | Patients: Behavioral Activation Therapy (BA)
Number analyzed (Participants) | 208 | 208
Participants
  Total Number of Deaths at 3-months | 16 | 7
  Total Number of Deaths at 6-months | 24 | 15
  Total Number of Deaths at 12-months | 36 | 27
Statistical Analysis 1: Comparison: Patients: Medication Management (MEDS) vs Patients: Behavioral Activation Therapy (BA); Test type: Superiority; p > 0.05, Kaplan Meier survival plots — The a priori threshold for statistical significance is p<0.05

ADVERSE EVENTS:
Time Frame: 1 year
Description: We collected information about all-cause mortality, serious adverse events, and other adverse events, using a standardized data collection form and summary form where a description of the event was provided. All-cause mortality, serious adverse events, and other (not including serious) adverse events were not monitored/assessed for caregivers. Adverse events were monitored/assessed without regard to the specific adverse event term.
Groups:
- Patients: Medication Management (MEDS): The medication management group will meet with the patient in a one 50 minute in person introductory antidepressant medication treatment session to educate the patient about depression and medication options. Patients will get prescribed a standard of care anti-depressant medication by treating physician, followed by 12 weekly follow up telephone visits, then on a monthly basis for 3 months, and then as needed thereafter.
  Medication Management: Collaborative care model will be used. The medication management group will meet with the patient in a one 50 minute in person introductory antidepressant medication treatment session to educate the patient about depression and medication options. Patients will get prescribed a standard of care anti-depressant medication by treating physician, followed by 12 weekly follow up telephone visits, then on a monthly basis for 3 months, and then as needed thereafter.
  Caregivers did not receive active treatment, however they were assessed for caregiver burden using the Caregiver Burden Questionnaire at 3, 6, and 12 months.
- Patients: Behavioral Activation Therapy (BA): BA is an evidence-based psychotherapy with more than 25 randomized trials showing effectiveness in depression. The therapy group will consist of an introductory in person 50-minute treatment session, followed by 12 weekly telephone 50-minute outpatient treatment sessions, then 3 monthly telephone 50-minute outpatient maintenance sessions. A typical BA session will last 50 minutes and include a review of the previous session and completed daily monitoring record forms, an in-depth discussion of life areas and value, and verbal reinforcement of activity engagement.
  Behavioral Activation Therapy: The therapy group will consist of an introductory in person 50-minute treatment session, followed by 12 weekly telephone 50-minute outpatient treatment sessions, then 3 monthly telephone 50-minute outpatient maintenance sessions. A typical BA session will last 50 minutes and include a review of the previous session and completed daily monitoring record forms, an in-depth discussion of life areas and value, and verbal reinforcement of activity engagement.
  Caregivers did not receive active treatment, however they were assessed for caregiver burden using the Caregiver Burden Questionnaire at 3, 6, and 12 months.
Arm/Group | Patients: Medication Management (MEDS) | Patients: Behavioral Activation Therapy (BA)
All-Cause Mortality (participants affected / at risk) | 36/208 | 27/208
Serious Adverse Events (participants affected / at risk) | 36/208 | 27/208
Other Adverse Events (participants affected / at risk) | 0/208 | 0/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients: Medication Management (MEDS) (N=208) | Patients: Behavioral Activation Therapy (BA) (N=208)
All-Cause Mortality (General disorders) | 36 (36) | 27 (27) — Deemed by DSMB as not related to study interventions.

LIMITATIONS AND CAVEATS:
For our secondary outcomes of Emergency Department Visits, Hospital Readmissions, and Total Days in the Hospital, we were only able to collect such data for ED visits and hospital admissions that occurred at Cedars-Sinai Medical Center and outside institutions that share data with the Cedars-Sinai Health System. As such, this data may not be complete since patients could potentially have visited different hospitals that we do not know about.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/00/NCT03688100/Prot_SAP_000.pdf